CLINICAL TRIAL: NCT05289635
Title: Effect of Different Suture Techniques on Early Healing of Peri-implant Soft Tissue Following Open-flap Implant Surgery in Esthetic Area: a Randomized Clinical Trial Comparing Horizontal and Vertical Mattress Sutures
Brief Title: Effect of Different Suture Techniques on Early Healing of Peri-implant Soft Tissue
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Junyu Shi, Dr., Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SH9th-03-07
Record Dates: First submitted 2022-03-06; First posted 2022-03-21 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Dental Implants; Wound Healing; Sutures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental): vertical mattress suture
  Interventions: Procedure: different suture types
- control group (Other): horizontal mattress suture
  Interventions: Procedure: different suture types

INTERVENTIONS:
Procedure: different suture types — For a wound that is deeper in nature, a mattress stitch can be placed, providing better strength. Mattress sutures can be applied as vertical or horizontal subtypes. So far, various studies have compared the effect of horizontal mattress suture (HMS) with vertical mattress suture (VMS) on wound healing in different wound. However, limited studies have evaluated the effect of the subtype of mattress sutures on the early wound healing and microcirculation changes of peri-implant soft tissues following implant surgery using Laser Doppler flowmetry. The test group use vertical mattress suture and the control group use the horizontal mattress suture.

SUMMARY:
The purposes of this study are to compare the blood perfusion and early healing of horizontal mattress suture with vertical mattress sutures following open-flap implant surgery. Patients wanting single implant replacement in esthetic area will be recruited. This is a randomized, open-label, controlled clinical trial. Noninvasive procedures will be used to assess the primary and secondary outcomes.

Inclusion Criteria: With sufficient bone width (≥6mm), With mesial-distal distance over 8mm, age over 18, Willing to participate Exclusion Criteria: Patients want multiple adjacent implant replacements in esthetic area, Untreated periodontitis, Smokers, Diabetes mellitus

DETAILED DESCRIPTION:
The overall aim of this study is to compare the microcirculation changes of peri-implant soft tissues following open-flap implant surgery using different suture techniques. Subjects fulfilling the inclusion and exclusion criteria will be invited to participate in the study and randomized to one of the two groups: vertical mattress suture (test group) and horizontal mattress suture (control group) on a 1:1 ratio. A laser Doppler flowmetry machine (LDF) (LW1111, LEA) will be used to measure the tissue perfusion. Assessment will be performed at different time, including: Baseline Assessments (presurgical measurements) - T0; Immediate after anesthesia - T1; Immediate after suture - T2; 1 hour after surgery - T3; 2 hours after surgery - T4; 6 hours after surgery - T5; 24 hours after surgery - T6; 72 hours after surgery - T7; 7 days after surgery - T8; 14 days after surgery - T9; 30 days after surgery - T10. The primary outcome is blood perfusion volume (PU) change during the observation period. And secondary outcomes include blood flow velocity change during the observation period, hemoglobin count change during the observation period, blood oxygen saturation change during the observation period; three-dimensional soft-tissue volumetric changes during the observation period, changes in clinical wound healing score during the observation period, PROMs (VAS).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 and above
2. Subjects want single implant treatment in esthetic area (premolar to premolar) in maxilla
3. With sufficient bone width (≥6mm)
4. With mesial-distal distance over 8mm
5. Evidence of subject ability to achieve good oral hygiene and control periodontitis in the whole of the dentition (FMPS<20% and FMBS<20%)
6. Ability to understand study procedures and to comply with them for the entire length of the study. Ability and willingness to give written informed consent.

Exclusion Criteria:

1. Subjects want multiple adjacent implant treatment
2. Patients with inadequate bone volume where major bone augmentation would be required at implant location.
3. Subjects with untreated periodontitis
4. Current smokers
5. Subjects with diabetes mellitus.
6. Pregnant females
7. Participation in another intervention trial
8. Inability or unwillingness of individual to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Blood perfusion volume (PU) change during the observation period | Immediate after anesthesia;Immediate after suture;1hour after surgery;2hour after surgery;6hour after surgery;24hour after surgery;72hour after surgery;7days after surgery;14ddays after surgery;30days after surgery
  LEA measurement

SECONDARY OUTCOMES:
Blood flow velocity change during the observation period | Immediate after anesthesia;Immediate after suture;1 hour after surgery;2hour after surgery;6hour after surgery;24hour after surgery;72hour after surgery;7 days after surgery;14days after surgery;30days after surgery
  LEA measurement
Hemoglobin count change during the observation period | Immediate after anesthesia;Immediate after suture;1 hour after surgery;2hour after surgery;6hour after surgery;24hour after surgery;72hour after surgery;7 days after surgery;14days after surgery;30days after surgery
  LEA measurement
Blood oxygen saturation change during the observation period | Immediate after anesthesia;Immediate after suture;1 hour after surgery;2hour after surgery;6hour after surgery;24hour after surgery;72hour after surgery;7 days after surgery;14days after surgery;30days after surgery
  LEA measurement
Three-dimensional soft-tissue volumetric changes during the observation period | 1. Intra-oral scanning: before surgery;Immediate after suture;1 hour after surgery;2hour after surgery;6hour after surgery;24hour after surgery;72hour after surgery;7 days after surgery;14days after surgery;30 day after surgery
  Intra-oral scanning; the thickness of the soft tissue
Changes in clinical wound healing score during the observation period | 24h after surgery;72h after surgery;7 days after surgery;14days after surgery;30 days after surgery
  Clinical measurements and clinical photographs. A modified healing index (Masse 1993)
  1. tissue color (1 = the gingival tissue was entirely pink; 2 = less than half of the gingival tissue was red, movable, and hyperemic;3 = more than half of the gingival tissue was red, movable, and hyperemic)
  2. healing tissue consistency and color (l=pink, close-grained; 2=red, soft; 3=gray-green, fragile)
  3. bleeding (l= none; 2=only upon palpation; 3=spontaneous) suppuration (1= none; 2=none, but significant amounts of plaque around the walls of the socket; 3=suppuration.
patient reported outcome measures (PROMs, VAS) | Immediate after suture;6hour after surgery;24hour after surgery;72hour after surgery;7 days after surgery;
  A horizontal line about 10 cm long was used, with "0" and "10" ends at each end, with 0 being no pain and 10 being the most severe pain that was unbearable.
  Visual analogue scale (0-10) will be used to evaluate the post-operative pain.

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio S. Tonetti, Professor, Study Chair — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Marsidi N, Vermeulen SAM, Horeman T, Genders RE. Measuring Forces in Suture Techniques for Wound Closure. J Surg Res. 2020 Nov;255:135-143. doi: 10.1016/j.jss.2020.05.033. Epub 2020 Jun 16. PMID 32543379
- [Result] Montanez A, Makarewich CA, Burks RT, Henninger HB. The Medial Stitch in Transosseous-Equivalent Rotator Cuff Repair: Vertical or Horizontal Mattress? Am J Sports Med. 2016 Sep;44(9):2225-30. doi: 10.1177/0363546516648680. Epub 2016 Jun 8. PMID 27281277
- [Result] Maemura K, Mataki Y, Kurahara H, Tanoue K, Kawasaki Y, Ijichi T, Iino S, Ueno S, Shinchi H, Natsugoe S. The 1-year outcomes after pancreaticogastrostomy using vertical versus horizontal mattress suturing for gastric wrapping. Surg Today. 2021 Apr;51(4):511-519. doi: 10.1007/s00595-020-02134-z. Epub 2020 Sep 23. PMID 32968859
- [Result] Wachtel H, Schenk G, Bohm S, Weng D, Zuhr O, Hurzeler MB. Microsurgical access flap and enamel matrix derivative for the treatment of periodontal intrabony defects: a controlled clinical study. J Clin Periodontol. 2003 Jun;30(6):496-504. doi: 10.1034/j.1600-051x.2003.00013.x. PMID 12795787
- [Result] Burkhardt R, Lang NP. Role of flap tension in primary wound closure of mucoperiosteal flaps: a prospective cohort study. Clin Oral Implants Res. 2010 Jan;21(1):50-4. doi: 10.1111/j.1600-0501.2009.01829.x. PMID 20070747

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT05289635/Prot_SAP_000.pdf